CLINICAL TRIAL: NCT02941627
Title: The Neuro Zti Cochlear Implant System Efficacy and Safety in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIC_07
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Cochlear; Deafness
Keywords: Hearing Loss; Cochlear Implant surgery; Otorhinolaryngology; Oticon Medical; Neuro Cochlear Implant System
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuro Cochlear Implant System study group (Experimental): All patients will receive a Neuro Zti implant and fitted with Neuro One sound processor
  Interventions: Device: Neuro Zti; Device: Neuro One

INTERVENTIONS:
Device: Neuro Zti — Cochlear implant
Device: Neuro One — Sound processor

SUMMARY:
The purpose of the study is to assess the efficacy and the safety profile of the Neuro Cochlear Implant System (CIS) in adults with severe-to-profound hearing loss.

DETAILED DESCRIPTION:
Appropriate adult cochlear implant candidates with sensorineural hearing loss, from English French Canadian centres and Danish centre, received Neuro Zti cochlear implant and fit with Neuro One sound processor.

Speech perception testing, using HINT (Hearing In Noise Test) sentences in quiet (65 dB SPL) (decibel, Sound Pressure Level) and in noise (+10 dB SNR) (decibel, Signal-to-Noise-Ratio), will be administrated pre-operatively in the best listening conditions and 3, 6, and 12 months post-activation in the implanted ear.

Adverse events will be collected during the surgery and over the post-surgical period from activation to12 months post-activation.

Safety will be assessed on the overall English, French and Danish participants. Efficacy will be assessed on English speaking participants.

ELIGIBILITY:
Inclusion criteria

* Adults, eighteen (18) years of age or older.
* Bilateral severe-to-profound sensorineural hearing loss, defined by pure-tone average (PTA) ≥70 dB HL (Hearing Level) at 500, 1000 and 2000 Hz on both ears.
* HINT sentences recognition scores in quiet ≤ 50% correct, in the best-aided listening condition.
* Post-lingual onset of deafness.
* Primary implantation (no re-implantation).
* Up-to-date pneumococcal vaccine.

Exclusion criteria

* Medical conditions that contraindicate undergoing cochlear implant surgery (middle ear diseases i.e. AOM/CSOM (Acute Otitis Media/Chronic Suppurative Otitis Media) , lesions of auditory nerve, pathologies of central auditory pathway, otosclerosis; cochlear malformation i.e. Mondini malformation, cochlear ossification, large vestibular aqueduct).
* Unrealistic expectations regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and medical device.
* Unwillingness or inability of the candidate to comply with all investigational requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schramm, MD, Principal Investigator — Ottawa Civic Hospital; Daniel Philippon, MD, Principal Investigator — CHU de Quebec; Joseph Chen, MD, Principal Investigator — Sunnybrook Hospital -Toronto; Nael Shoman, MD, Principal Investigator — Royal University Hospital, Saskatoon; David P. Morris, MD, Principal Investigator — Nova Scotia Hearing and Speech Centres - Halifax; Per Cayé Thomasen, MD, Principal Investigator — Gentofte Hospital
Locations (6):
- Canada (5):
  - Nova Scotia Hearing and Speech centres, Halifax
  - Ottawa Civic Hospital, Ottawa
  - CHU de Quebec - Université de Laval, Québec
  - Royal University Hospital, Saskatoon
  - Sunnybrook Hopital, Toronto
- Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The present clinical trial started enrolling in Feb. 2017, therefore it does not contain a data sharing statement or Individual Participant Data sharing statement. Data will be analyzed as patient group data and submitted for peer-reviewed publication.

REFERENCES:
- [Result] Schramm D, Chen J, Morris DP, Shoman N, Philippon D, Caye-Thomasen P, Hoen M, Karoui C, Laplante-Levesque A, Gnansia D. Clinical efficiency and safety of the oticon medical neuro cochlear implant system: a multicenter prospective longitudinal study. Expert Rev Med Devices. 2020 Sep;17(9):959-967. doi: 10.1080/17434440.2020.1814741. Epub 2020 Oct 3. PMID 32885711
- See also: oticon medical website — https://www.oticonmedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Efficacy outcomes will be based on English speaking participants, and safety on overall patients; English, French and Danish speaking participants.
Groups:
- Neuro Zti/Neuro One Study Group: All patient will receive a Neuro Zti implant and fit with Neuro One sound processor.
Period: Overall Study
Arm/Group | Neuro Zti/Neuro One Study Group
Started | 53 (Among 53 patients enrolled: 1 passed away after the informed consent completion, 1 was not implanted for surgical failure, and 1 for cholesteatoma discovered during surgical procedure. This last patient was included in safety analysis as defined in the protocol. Therefore, among 53 patients enrolled 51 were evaluated for safety outcomes, and 50 were successfully implanted and complete the study.)
Clinical Safety on Overall Participants | 51
Clinical Efficiency on English Speaking Participants | 33 (Among the 50 patients successfully implanted 33 English speaking participant complete speech performance measure.)
Completed | 50
Not Completed | 3
Not completed — Death | 1
Not completed — Surgical failure | 1
Not completed — cholesteatoma prevented implantation | 1

BASELINE CHARACTERISTICS:
Population: Fifty-one (51) participants with post-lingual severe-to-profound hearing loss took part in the study. One (1) subject could not be implanted because of the discovery during surgery of cholesteatoma (i.e., keratinized tissue growth in the middle ear or mastoid process) that was not detected before. The cochlear implantation was converted into choleastoma removal surgery.
Groups:
- Neuro Zti/Neuro One Study Group: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients will receive a Neuro Zti implant and fit with Neuro One sound processor
Arm/Group | Neuro Zti/Neuro One Study Group
Number analyzed (Participants) | 51
Age, Customized [Count of Participants; unit: Participants]
  [18;40] years old | 1
  [40;50] years old | 2
  [50;60] years old | 7
  >=60 years old | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Age at implantation [Mean (Standard Deviation); unit: years] | 69.5 (11.4)
Primary hearing loss etiology [Count of Participants; unit: Participants]
  Aging | 3
  Genetics | 7
  Noise exposure | 7
  Menière's disease | 3
  Other | 6
  Unknown | 23
  Otosclerosis | 1
  Viral | 1
Implanted ear (side) [Number; unit: participants]
  Left | 22
  Right | 29
Duration of hearing loss [Mean (Standard Deviation); unit: years]
  Implanted ear | 30.7 (19.0)
  Contralateral ear | 33.2 (19.6)
Duration of hearing aid use [Mean (Standard Deviation); unit: years]
  Implanted ear | 22.2 (15.8)
  Contralateral ear | 22.6 (15.8)
PTA (Pure Tone Average), 500 Hz to 2000 Hz [Mean (Standard Deviation); unit: dB HL]
  Implanted ear | 101.3 (13.3)
  Contralateral ear | 95.8 (16.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing In Noise Test Score in Quiet (HINT-Q) From Baseline to 6 Months in English-speaking Participants.
Description: To assess the clinical efficiency, speech perception performance using the HINT sentences was measured in quiet at 6 months pos-activation in English speaking participants.
  Primary clinical efficiency outcome is defined as the change in HINT scores from baseline to 6 months post-activation.
  Recorded HINT sentences lists were presented to the participant at 60 dB SPL (sound pressure level) pre-operatively in the best aided hearing conditions and at 6 months in the implanted ear after Neuro Zti implant activation. The post-activation assessment was performed in the implanted ear alone with masked controlateral ear. Resultant score is a percentage of words correctly repeated. Possible scores are range from 0% to 100% words correctly repeated. Change = (6 Months score - Baseline score). A score greater or equal to 10% was considered clinically significant improvement.
Time Frame: pre-operative, 6 Months
Population: Clinical efficiency is reported on the thirty-three (33) English-speaking participants.
Measure: Mean (Standard Deviation); unit: percent change words correctly repeated
Groups:
- Neuro Zti/Neuro One English-Speaking Participants - 6 Months: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor
Arm/Group | Neuro Zti/Neuro One English-Speaking Participants - 6 Months
Number analyzed (Participants) | 33
percent change words correctly repeated | 51.5 (33.1)

2. Primary Outcome: Major Related Adverse Event (AE)
Description: Adverse event (AE) is defined as any undesired change from the participant's baseline condition symptom or clinically relevant symptom or disease, regardless of its cause.
  AEs include complications that are related to the device or clinical procedure, as well as unrelated AE that are not related to the device or the trial procedure.
  AEs were classified as Major if they corresponded to any of the following criteria:
  * life-threatening conditions (e.g. meningitis)
  * require hospitalization
  * result in permanent disability or damage (e.g. facial nerve paresis)
  * require revision surgery with or without explantation or re-implantation (e.g. device failure, flap necrosis)
  * medical events that could not be alleviated by electrode deactivation (e.g. tinnitus, facial nerve stimulation, pain)
  The co-primary safety endpoint is the major related adverse events rate during the surgery and over the post-surgical period from activation to 12 months post-activation.
Time Frame: 12 months
Population: Safety is reported, on overall participants, in terms of surgical safety (intra-operative major complication rate) and post-surgical safety (major complication rate from the surgery to 12 months post activation to determine the long-term safety profile of the Neuro cochlear implant system).
Measure: Number; unit: number of major adverse events
Units Other Than Participants: number of adverse events
Groups:
- Neuro Zti/Neuro One Study Group: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor.
Arm/Group | Neuro Zti/Neuro One Study Group
Number analyzed (Participants) | 51
Number analyzed (number of adverse events) | 71
number of major adverse events
  Major device related AE: number analyzed (number of adverse events) | 1
  Major device related AE | 1
  Major trial procedure related AE: number analyzed (number of adverse events) | 1
  Major trial procedure related AE | 1
  Major unrelated AE: number analyzed (number of adverse events) | 2
  Major unrelated AE | 2

3. Secondary Outcome: Clinical Benefit on English-speaking Participants
Description: Clinical benefit is defined as the change of HINT scores post-operatively in the implanted ear only with masked contralateral ear and pre-operatively in the best aided conditions. Clinical benefit is measured in quiet and in noise using the Hearing in Noise Test (HINT).
  In quiet, HINT sentences lists were presented to the participant at 60 decibel sound pressure level (dB SPL). In noise, the sentences were presented with concurrent background noise at +10 decibel signal-to-noise-ratio (dB SNR), signal level at 65 dB SPL and noise at 55 dB SPL. Resultant score is a percentage of words correctly repeated, possibly ranged from 0% to 100%.
  Clinical benefit is computed for each participant. A positive difference of post- and pre-operative HINT scores is considered clinically significant if it exceeded 10 percentage points (pp). A decrease that exceeded 10 pp is considered a clinically significant decrement. A difference of less than 10 pp was considered as no change in performance.
Time Frame: 3, 6 and 12 months
Population: Clinical benefit is reported on the English-speaking participants.
Measure: Count of Participants; unit: Participants
Groups:
- Neuro Zti/Neuro One English-speaking Participants 3 Months: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor
  Clinical benefit is assessed in English-speaking participants at 3 months follow up.
- Neuro Zti/Neuro One English-speaking Participants 6 Months: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor
  Clinical benefit is assessed in English-speaking participants at 6 months follow-up
- Neuro Zti/Neuro One English-speaking Participants 12 Months: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor
  Clinical benefit is assessed in English-speaking participants at 12 months follow-up
Arm/Group | Neuro Zti/Neuro One English-speaking Participants 3 Months | Neuro Zti/Neuro One English-speaking Participants 6 Months | Neuro Zti/Neuro One English-speaking Participants 12 Months
Number analyzed (Participants) | 33 | 33 | 33
Participants
  HINT sentences in Quiet (60dB SPL): Better (> 10 percent points) | 26 | 29 | 30
  HINT sentences in Quiet (60dB SPL): Similar (-10 to 10 percent points) | 2 | 3 | 2
  HINT sentences in Quiet (60dB SPL): Worse (< -10 percent points) | 5 | 1 | 1
  HINT sentences in Noise (+10 dB SNR): Better (> 10 percent points) | 22 | 24 | 27
  HINT sentences in Noise (+10 dB SNR): Similar (-10 to 10 percent points) | 7 | 6 | 6
  HINT sentences in Noise (+10 dB SNR): Worse (< -10 percent points) | 4 | 3 | 0

4. Secondary Outcome: Hearing In Noise Test Score in Quiet (HINT-Q) Pre-operatively, at 3-, 6- and 12-Months on English-speaking Participants
Description: To assess the clinical efficiency, speech perception performance using the HINT sentences was measured in quiet pre-operatively, 3-, 6- and 12-months pos-activation on English speaking participants.
  Secondary clinical efficiency outcome is defined as the mean HINT scores from baseline to 12 months post-activation.
  Recorded HINT sentences lists were presented to the participant at 60 dB SPL pre-operatively in the best aided hearing conditions, at -, 6- and 12- months. The post-activation assessment was performed in the implanted ear alone with masked controlateral ear. Resultant score is a percentage of words correctly repeated. Possible scores are range from 0% to 100% words correctly repeated. A higher score is better.
Time Frame: pre-operative, 3, 6 and 12 Months
Population: Clinical efficiency is reported on the thirty-three (33) English-speaking participants.
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Groups:
- Neuro Zti/Neuro One English Speaking Participants: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor
Arm/Group | Neuro Zti/Neuro One English Speaking Participants
Number analyzed (Participants) | 33
percentage of words correctly repeated
  HINT-Q score at baseline in best aided conditions | 13.3 (16.0)
  HINT-Q score at 3 months in implanted ear | 55.8 (31.8)
  HINT-Q score at 6 months in implanted ear | 64.8 (27.2)
  HINT-Q score at 12 months in implanted ear | 70.1 (24.5)

5. Secondary Outcome: Hearing In Noise Test Score in Noise (HINT-N) Pre-operatively, at 3-, 6- and 12-Months on English-speaking Participants
Description: To assess the clinical efficiency, speech perception performance using the HINT sentences was measured in noise pre-operatively, 3-, 6- and 12-months pos-activation on English speaking participants.
  Secondary clinical efficiency outcome is defined as the mean HINT scores from baseline to 12 months post-activation.
  Testing open-set sentence recognition with concurrent background noise present at +10 decibel signal-to-ratio (dB SNR) with signal level presented at 65 dB SPL and noise at 55 dB SPL. Recorded HINT sentences lists were presented to the participant in front pre-operatively in the best aided condition and post-operatively in the implanted ear alone with masked contralateral ear. Speech and noise were colocated (S0N0). Resultant score is a percentage of words correct. Possible scores range from 0% to 100% words correctly repeated. A higher score is better.
Time Frame: pre-operative, 3-, 6- and 12-Months
Population: Clinical efficiency is reported on the thirty-three (33) English-speaking participants.
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Arm/Group | Neuro Zti/Neuro One English Speaking Participants
Number analyzed (Participants) | 33
percentage of words correctly repeated
  HINT-N score at baseline in best aided condition | 13.3 (17.7)
  HINT-N score at 3 months in implanted ear | 43.8 (30.6)
  HINT-N score at 6 months in implanted ear | 52.3 (30.0)
  HINT-N score at 12 months in implanted ear | 57.6 (29.9)

6. Secondary Outcome: Minor Adverse Events (AE)
Description: Adverse event (AE) is defined as any undesired change from the participant's baseline condition symptom or clinically relevant symptom or disease, regardless of its cause.
  AEs include complications that are related to the device or clinical procedure, as well as unrelated AE that are not related to the device or the trial procedure.
  AEs were classified as Minor if they corresponded to any of the following criteria:
  * adverse event settled spontaneously without surgical procedure (e.g. hematoma)
  * adverse event settled spontaneously with conservative medical management
  The secondary safety endpoint is the minor related adverse events rate during the surgery and over the post-surgical period from activation to 12 months post-activation.
Time Frame: 12 months
Population: Safety is reported, on overall participants, in terms of surgical safety (intra-operative minor complication rate) and post-surgical safety (minor complication rate from the surgery to 12 months post activation to determine the long-term safety profile of the Neuro cochlear implant system).
Measure: Number; unit: number of minor adverse events
Units Other Than Participants: number of adverse events
Groups:
- Overall Study Participants: Neuro Zti: cochlear implant Neuro One: sound processor
  All patients received a Neuro Zti implant and fitted with Neuro One sound processor
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 51
Number analyzed (number of adverse events) | 71
number of minor adverse events
  Device related AE | 16
  Trial procedure related AE | 20
  Unrelated AE | 31

ADVERSE EVENTS:
Time Frame: From the participant's cochlear implant surgery initiation to the end of month 12.
Description: Safety Analysis was based on participants for whom the surgery for cochlear implantation was initiated. Among 53 patients enrolled: 1 died for heart stroke after the informed consent process, 1 was not implanted for surgical failure, and 1 for cholesteatoma discovered during surgical procedure. This patient was included in safety analysis as defined in the protocol. Then, among 53 patients enrolled 51 were evaluated for safety outcomes, 50 were successfully implanted and complete the study.
Groups:
- Neuro Zti/Neuro One Study Group: Neuro Zti: implant Neuro One: sound processor All patient will receive a Neuro Zti implant and fit with Neuro One sound processor.
Arm/Group | Neuro Zti/Neuro One Study Group
All-Cause Mortality (participants affected / at risk) | 1/53
Serious Adverse Events (participants affected / at risk) | 3/51
Other Adverse Events (participants affected / at risk) | 15/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neuro Zti/Neuro One Study Group (N=51)
Diagnosis of Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Hepatic cancer
Kidney failure (Renal and urinary disorders) | 1
Exacerbation of COPD (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neuro Zti/Neuro One Study Group (N=51)
Tinnitus (Ear and labyrinth disorders) | 4
Post operative dizziness (Injury, poisoning and procedural complications) | 8
Post procedural pain (Injury, poisoning and procedural complications) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No independent manuscript is submitted for publication until the multicentre manuscript is accepted for publication. PI can publish results from his/her own site after multicentre manuscript is accepted for publication or 18 months after study completion. Independent manuscript must be submitted to Sponsor for review at least 30 days prior to publication. Sponsor can request within the 30-day review period, PI shall delay proposed communication up to 60 days from the date of Sponsor's request.

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT02941627/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT02941627/SAP_001.pdf